CLINICAL TRIAL: NCT07333950
Title: The Efficacy and Safety of Endovascular Therapy for Acute Ischemic Stroke Due to Large Core Infarction -- A Multicenter, Prospective, Open-label, Blind Endpoint, Randomized Controlled Trial
Brief Title: The Efficacy and Safety of Endovascular Therapy for Acute Ischemic Stroke Due to Large Core Infarction
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Feng Gao, Vice-Director of Interventional Neuroradiology, Department of Neurology, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HX-A-2025081
Record Dates: First submitted 2025-12-22; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Acute Basilar Artery Occlusion; Endovascular Therapy; Large Core Infarction
Keywords: Ischemic Stroke; Acute Basilar Artery Occlusion; Endovascular Therapy; Large Core Infarction
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endovascular Treatment Group (Experimental): Participants randomized to the endovascular recanalization arm will receive endovascular treatment in addition to best medical management. The procedure aims to achieve recanalization of the occluded posterior circulation vessel using mechanical thrombectomy techniques, including stent retriever and/or aspiration-based approaches. When necessary, adjunctive endovascular measures may be performed as rescue therapy at the discretion of the treating neurointerventionalist.
  Interventions: Procedure: Endovascular Recanalization Strategy
- Best Medical Management Group (Other): Participants randomized to this arm will receive best medical management alone, consistent with current guideline recommendations for the acute and secondary prevention phases of ischemic stroke. No endovascular recanalization procedures are permitted after randomization.
  Interventions: Drug: Best Medical Management

INTERVENTIONS:
Procedure: Endovascular Recanalization Strategy — The endovascular approach is selected by the treating neurointerventionalist based on angiographic findings, occlusion characteristics, and procedural feasibility. Permitted techniques include mechanical thrombectomy using stent retriever and/or aspiration-based methods. Adjunctive endovascular procedures, such as balloon angioplasty, stent placement, or intra-arterial thrombolysis, may be used when deemed necessary to achieve or maintain vessel patency. Angiographic reperfusion is assessed during the procedure, and treatment is terminated once adequate revascularization is obtained. Subsequent medical management is individualized according to stroke mechanism, procedural findings, and post-treatment imaging.
  Arms: Endovascular Treatment Group
Drug: Best Medical Management — Best medical management consists of comprehensive evidence-based medical therapy for acute ischemic stroke, encompassing acute supportive care, neurological and physiological monitoring, etiological evaluation, and secondary prevention strategies. Standard pharmacological treatments are administered as appropriate, together with risk factor modification and supportive care measures, in accordance with current guideline recommendations. Endovascular recanalization procedures are not included in this treatment strategy.
  Arms: Best Medical Management Group

SUMMARY:
This study assesses the efficacy and safety of endovascular therapy in patients with acute basilar artery occlusion with large core infarction within a multicenter, prospective, open-label, blinded endpoint, randomized controlled trial

DETAILED DESCRIPTION:
This is a prospective, randomized, open-label, controlled trial designed to compare 90-day clinical outcomes between endovascular therapy (EVT) and best medical management (BMM) in patients with acute posterior circulation large vessel occlusion (LVO) and large core infarction. Eligible patients, aged 18 to 80 years presenting within 24 hours of symptom onset or last known well, must have imaging-confirmed acute basilar artery occlusion and large core infarction, defined as a pc-ASPECTS ≤5 or a Pons-midbrain-index (PMI) ≥ 3 on NCCT or DWI. Participants will be randomly assigned (1:1) to receive EVT or BMM. The primary outcome is functional independence at 90 days, assessed by the proportion of patients achieving a modified Rankin Scale (mRS) score of 0-3. Secondary outcomes include the distribution of mRS scores at 90 days, 90-day all-cause mortality, and the incidence of symptomatic intracranial hemorrhage (sICH)

ELIGIBILITY:
Inclusion Criteria:

1. The age ranged from 18 to 80 years
2. Acute ischemic stroke in posterior circulation, the time from stroke onset (or finally found normal) to randomization was within 24 hours
3. Acute basilar artery occlusion confirmed by CTA,MRA,or DSA
4. Posterior circulation large core infarction:NCCT or DWI showed pc-ASPECTS≤5, or Pons-Midbrain Index (PMI)≥3
5. NIHSS score ≥10 before randomization
6. Pre-stroke mRS of 0-2
7. Each patient or their legal representative must provide written informed consent before enrolment

Exclusion Criteria:

1. Any sign of intracranial hemorrhage (except microbleeds) on brain imaging prior to randomization
2. Complete cerebellar infarct with significant mass effect, or bilateral thalamic infarction as evidenced by baseline neuroimaging
3. Known or highly suspected chronic occlusion of basilar artery
4. History of contraindication for contrast medium (except mild rash)
5. Current pregnant or breast-feeding
6. Refractory hypertension (defined as systolic blood pressure>220 mmHg or diastolic blood pressure>110 mmHg) that cannot be controlled by drug treatment;
7. Known to have dementia or psychiatric disease unable to complete neurological assessment and follow-up
8. It is known that patients with dementia or mental illness cannot complete neurological function assessment and follow-up
9. Patients whose life expectancy is less than 1 year (such as patients with malignant tumor, advanced cardiopulmonary disease, etc.)
10. Enrolled in another drug or device trial or expected to participate in another drug or device treatment trial within the following 3 months
11. Any other condition (in the opinion of the site investigator) that inappropriate to participate this study
12. CTA/MRA/DSA confirmed occlusion of anterior and posterior circulation
13. Central nervous system vasculitis has been diagnosed or clinically suspected
14. Known hereditary or acquired bleeding tendency, lack of coagulation factors, or oral anticoagulants with INR>1.7
15. Blood glucose<2.7 or>22.2 mmol/L; Platelet count<50×109/L, glomerular filtration rate<30ml/min or serum creatinine ≥ 3 mg/dl
16. Acute cerebral infarction occurred within 48 hours after cardio cerebral vascular intervention or major surgery (patients over 48 hours can be included in the group)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 308 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of modified Rankin scale 0-3 at 90 (±14) days after randomization | 90±14 days after randomization
  The modified Rankin scale (mRS) ranged from 0 to 6, with a score of 0 indicating no disability, 1 no clinically significant disability, 2 slight disability, 3 moderate disability but remaining able to walk unassisted, 4 moderately severe disability,5 severe disability, and 6 death.

SECONDARY OUTCOMES:
MRS score as an ordinal scale at 90 (±14) days after randomization | 90±14 days after randomization
  The modified Rankin scale (mRS) ranged from 0 to 6, with a score of 0 indicating no disability, 1 no clinically significant disability, 2 slight disability, 3 moderate disability but remaining able to walk unassisted, 4 moderately severe disability, 5 severe disability, and 6 death.
Rate of mRS 0-2 at 90 (±14) days after randomization | 90±14 days after randomization
  The modified Rankin scale (mRS) ranged from 0 to 6, with a score of 0 indicating no disability, 1 no clinically significant disability, 2 slight disability, 3 moderate disability but remaining able to walk unassisted, 4 moderately severe disability, 5 severe disability, and 6 death.
National Institutes of Health Stroke Scale (NIHSS) score at 24 hours after randomization | 24 hours after randomization
  The National Institute of Health Stroke Scale（NIHSS） ranged from 0 to 42, with higher scores indicating greater neurologic deficits.
NIHSS score at 7 days after randomization or discharge (whichever came first) | 7 days after randomization or at discharge
  The National Institute of Health Stroke Scale（NIHSS） ranged from 0 to 42, with higher scores indicating greater neurologic deficits.
Functional health status and quality of life (EuroQol Five Dimensions) at 90 (±14) days after randomization | 90±14 days after randomization
  EuroQol Five Dimensions (EQ-5D) is a standardized instrument for measuring the general health status. Rated level can be coded as a number 1, 2, 3, 4 or 5, which indicates having no problems for 1, having some problems for 2, having moderate problems for 3, having serious problems for 4 and having extreme problems for 5.
The proportion of Barthel Index ≥ 95 at 90 (± 14) days after randomization | 90±14 days after randomization
  The proportion of Barthel Index ≥ 95 at 90 (± 14) days after randomization.
Basilar artery recanalization at 18-36 hours after randomization (confirmed by CTA, MRA, DSA or TCD) | 18-36 hours after randomization
  Basilar artery recanalization at 18-36 hours after randomization (confirmed by CTA, MRA, DSA or TCD).
Technical success rate, defined as successful recanalization of target vessels at the end of surgery (eTICI 2b-3) | At the end of the operation
  Technical success rate, defined as successful recanalization of target vessels at the end of surgery (eTICI 2b-3).
The proportion of mRS 0-4 at 90 (± 14) days after randomization | 90±14 days after randomization
  The proportion of mRS 0-4 at 90 (± 14) days after randomization.

OTHER OUTCOMES:
Rate of any Symptomatic intracranial hemorrhage (sICH) defined as the Heidelberg classification within 18-36 hours of randomization | 18-36 hours after randomization
  Heidelberg standard was defined as new intracranial hemorrhage detected by brain imaging associated with any of the item below: 4 points total NIHSS at the time of diagnosis compared to immediately before worsening. 2 point in one NIHSS category. Leading to intubation/hemicraniectomy/ventricular drainage placement or other major medical/surgical intervention. Absence of alternative explanation for deterioration.
Rate of any intracranial hemorrhage identified by CT or MRI imaging within 18-36 hours after randomization | Any intracranial hemorrhage identified by CT or MRI imaging within 18-36 hours
  Any intracranial hemorrhage identified by CT or MRI imaging within 18-36 hours.
All cause of mortality within 7 days after randomization | 7 days after randomization
  All cause of mortality within 7 days after randomization
All cause of mortality within 90 (±14) days after randomization | 90±14 days after randomization
  All cause of mortality within 90 (±14) days after randomization

CONTACTS AND LOCATIONS:
Overall Officials: Feng Gao, MD, Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No